CLINICAL TRIAL: NCT06932783
Title: RESTORE: Remote Electrical Stimulation for Pain and Depression Treatment in Cirrhosis
Brief Title: Remote Electrical Stimulation for Pain and Depression Treatment in Cirrhosis
Acronym: RESTORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Elliot B. Tapper, Associate Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00269546
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Cirrhosis
Keywords: Transcutaneous Electrical Acustimulation; Chronic Pain; Depression
MeSH Terms: conditions — Fibrosis; Chronic Pain; Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to either TEA or sham-control. At least half of the participants will have depression per study definition.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Transcutaneous Electrical Acustimulation (TEA) (Experimental): Participants will have a two-week run-in period and then 8 weeks of treatment.
  Interventions: Device: Transcutaneous Electrical Acustimulation (TEA)
- TEA Sham (Sham Comparator): Participants will have a two-week run-in period and then 8 weeks of sham treatment.
  Interventions: Device: Sham Transcutaneous Electrical Acustimulation (TEA)

INTERVENTIONS:
Device: Transcutaneous Electrical Acustimulation (TEA) — Participant will apply TEA at home twice a day (approximately 45 minutes am/pm) for 8 weeks. The top electrode will be placed at ST36 (via acupuncture point) and the electrode patch will be placed vertically.
  Additionally, participants will agree to allow medical records to be collected, complete various surveys and have follow-up after treatment (approximately 9-10 weeks).
  Arms: Transcutaneous Electrical Acustimulation (TEA)
Device: Sham Transcutaneous Electrical Acustimulation (TEA) — Participant will apply sham TEA at home twice a day (approximately 45 minutes am/pm) for 8 weeks. Sham TEA will be performed via one point on the leg and not on any meridian or acupoints that were used in previous gastrointestinal studies and did not yield any significant effects.
  Additionally, participants will agree to allow medical records to be collected, complete various surveys and have follow-up after treatment (approximately 9-10 weeks)
  Arms: TEA Sham

SUMMARY:
This study is being done to better understand how the study team can treat pain for people with cirrhosis and depression.

Enrolled participants on this feasibility study will be randomized to Transcutaneous Electrical Acustimulation (TEA) or sham TEA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cirrhosis - must meet the criteria as outlined in the protocol
* Chronic pain (Patient self-reports ≥ 4 on the 0-10 scale for >50% of days within 3- months)
* Depression (in at least half of participants) - must meet the criteria as outlined in the protocol
* English speaking
* Willing to use a Transcutaneous Electrical Acustimulation device

Exclusion Criteria:

* Dementia and/or severe cognitive impairment
* Unable or unwilling to provide consent
* Expected to undergo liver transplant in next 24 weeks
* No email address
* Deemed unsuitable by the study investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Acceptability Questionnaire at 10 weeks | 10 weeks
  There are 7 questions that will be completed regarding the participant's experience with the study. There are six questions that participants will select strongly agree (5) - strongly disagree (1), with a range of 6-30. Additionally, participant's select from not very likely (1) -extremely likely (10).
  The last scale 1-10 asks "on a scale from 1-10, where 1 is not very likely and 10 is extremely likely, I am likely to recommend using the TEA device to a friend, colleague, or family member with cirrhosis and pain."
Feasibility based on the proportion of participants enrolled that were contacted | Enrollment period (2 years)
Feasibility based on the Proportion of enrolled participants that dropout (overall and during run in) | Run-in (-14 days to baseline) to 10 weeks
Feasibility based on time required to complete study assessments | Screening - 10 weeks
  Time will be in minutes
Proportion of questionnaires completed at baseline and the final study visit (10 weeks) | Baseline, 10 weeks
TEA usage during the intervention period | Weeks 1-8 of TEA treatment
  Time per day.

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Tapper, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No